CLINICAL TRIAL: NCT05124379
Title: Prospective, Open Clinical Investigation to Confirm the Effectiveness and Safety of Hemoclin Gel for the Treatment of Haemorrhoids.
Brief Title: Hemoclin Gel for the Treatment of Hemorrhoids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karo Pharma AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21E1799/HC_001
Record Dates: First submitted 2021-10-26; First posted 2021-11-18 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Hemorrhoids Grade I and II

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hemoclin Gel (Other)
  Interventions: Device: Hemoclin Gel

INTERVENTIONS:
Device: Hemoclin Gel — Non sterile gel for intra-rectal use

SUMMARY:
Post market, single arm, clinical investigation to assess safety and performance of the product.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects.
2. Sex: male or female.
3. Age: more than 18 years old.
4. Symptomatic haemorrhoids stage 1 and 2 (Goligher classification).
5. Episodes of haemorrhoid-related itching experienced at least every other day during the last two weeks before enrolment in the study.
6. Able to attempt bowel movements daily (defined as trying to have a bowel movement while sitting on the toilet for at least a few minutes, at least once daily, whether or not you feel the need to have a bowel movement that day).
7. Able and willing to provide informed consent and comply with study procedures

Exclusion Criteria:

1. Pregnant or nursing woman or planning a pregnancy during the study.
2. Subject not able or not willing to provide informed consent and comply with study procedures
3. Subject who had been deprived of their freedom by administrative or legal decision.
4. Major subject who is under guardianship or who is not able to express his consent.
5. Subject in a social or sanitary establishment.
6. Subject suspected to be non-compliant according to the Investigator's judgment. In terms of associated pathology
7. Grade III or IV haemorrhoids (Goligher classification).
8. Other pre-existing anal disorders and diseases including Crohns disease, ulcerative colitis, undefined inflammatory bowel disease, anal fissures, perianal fistulas, perianal rash or eczema, rectal prolapse, rectocele, benign or malignant anal and rectal tumor and perianal infections.
9. Any anal surgery (including surgical or instrumental procedures in the last 60 days). Relating to previous or ongoing treatment
10. Any anal topical medication applied in last 7 days.
11. Known or suspected sensitivity or allergy to ingredients of the investigational product. In terms of COVID pandemic
12. Subject who was abroad in a country with higher incidence rate of Covid-19 than Poland within 14 days before the beginning of the study.
13. Subject presenting following symptoms: cough, shortness of breath, elevated body temperature - equal and above 37.5°C.
14. Subject who had contact with any person infected with COVID-19 within 10 days before the beginning of the study.
15. Subject who is currently during home quarantine recommended by the Sanitary Inspection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2021-11-17 (Actual); Study Completion 2022-01-19 (Actual)

PRIMARY OUTCOMES:
The primary objective is to asses the treatment of itch related to Haemorrhoids grade I or II. | 2 weeks
  Severity of itch will be evaluated by the patient with a 6 point structured scale.

SECONDARY OUTCOMES:
To evaluate by the patient the efficacy of tested product on the severity of bleeding | 2 weeks
  Wilcoxon signed rank test will be carried out to assess whether the median change from baseline is statistically significant.
To evaluate by the patient the efficacy of tested product on the sense of discomfort | 2 weeks
  Wilcoxon signed rank test will be carried out to assess whether the median change from baseline is statistically significant.
To evaluate the overall satisfaction of the patient according to | 2 weeks
  Wilcoxon signed rank test will be carried out to assess whether the median change from baseline is statistically significant.
To evaluate the instant cooling effect, less painful toilet visit each day using a daily log, | 2 weeks
  Wilcoxon signed rank test will be carried out to assess whether the median change from baseline is statistically significant.

CONTACTS AND LOCATIONS:
Locations (1):
- GastroDent Gabinet Gastroenterologiczny z Pracownią Endoskopową", Gdansk, Poland

IPD SHARING:
Plan to Share IPD: No